CLINICAL TRIAL: NCT06552091
Title: Guided Digital Self-Hypnosis Solution for Managing Hot Flashes in Patients Undergoing Hormone Therapy
Acronym: HYBOU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-A01105-42
Record Dates: First submitted 2024-08-08; First posted 2024-08-13 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer Female
Keywords: breast cancer; non-metastatic; hormone therapy; hot flashes; self-hypnosis
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes

STUDY DESIGN:
Intervention Model Description: * Standard group: standard care.
  * Hypnosis group: experimental care with 3 self-hypnosis sessions over 3 weeks, one session per week to be practiced daily.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard group (No Intervention): standard care
- Hypnosis group (Experimental): experimental care with 3 self-hypnosis sessions over 3 weeks, one session per week to be practiced daily
  Interventions: Other: self-hypnosis sessions

INTERVENTIONS:
Other: self-hypnosis sessions — 3 self-hypnosis sessions over 3 weeks, one session per week to be practiced daily
  Arms: Hypnosis group

SUMMARY:
Patients treated for breast cancer with hormone therapy (HT) suffer from hot flashes. This side effect impacts treatment adherence. Indeed, approximately 50% of women take less than 80% of the prescribed dose, and up to 50% abandon their treatment before the fifth year of prescription, significantly increasing the risk of recurrence. Moreover, these hot flashes strongly impact the quality of life. According to the CANTO study, these hot flashes can persist up to two years after diagnosis, affecting social relationships, return to work, and physical and mental health.

Some side effects resulting from HT (sleep disturbances, fatigue, hot flashes) could be alleviated by a non-pharmacological approach involving the patient.

Our hypothesis is that a non-pharmacological solution, such as the use of self-hypnosis, could reduce hot flashes and the side effects related to HT or the perception thereof in patients treated for breast cancer. Consequently, this could improve the quality of life and lead to better treatment adherence.

The principal objective is to evaluate the effect of daily guided self-hypnosis sessions in reducing hot flashes in patients with non-metastatic breast cancer receiving anti-aromatase hormone therapy.

The secondary objectives are to evaluate :

* Patient adherence to guided self-hypnosis via a digital solution
* Quality of life
* Sleep quality
* Satisfaction with care
* Usability of the digital tool

The originality of this clinical trial is the proposal of self-hypnosis sessions over three weeks with three different themes using a digital solution.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient,
* WHO ≤ 2,
* Patient who is premenopausal, perimenopausal, or postmenopausal at diagnosis,
* Patient being treated for non-metastatic breast cancer,
* Ongoing adjuvant endocrine therapy, with or without concomitant anti-CDK 4/6 targeted therapy,
* Patient reporting at least 50 hot flashes per week or at least 7 hot flashes per day
* Patient has a computer device capable of accessing the self-hypnosis program link,
* Information provided and informed consent signed,
* Patient affiliated with the social security system.

Exclusion Criteria:

* Male,
* Patient with hearing impairments,
* Patient with psychotic and/or cognitive disorders As assessed by the clinician,
* Patient who does not understand the French language,
* Patient not diagnosed with non-metastatic breast cancer,
* Patient not undergoing anti-aromatase treatment,
* Patient reporting fewer than 50 hot flashes per week or fewer than 7 hot flashes per day,
* Prior participation in a hypnosis or self-hypnosis program before inclusion,
* Patient participating in a therapeutic program related to hot flashes,
* Patient already included in another therapeutic trial on the same topic,
* Patient already included in another therapeutic trial with an experimental drug,
* Pregnant or breastfeeding woman,
* Patient deprived of liberty (including guardianship and curatorship).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-02-17 (Estimated)

PRIMARY OUTCOMES:
Hot Flash Score (HFS) | 28 days
  In each group (standard and hypnosis), hot flashes will be primarily assessed using the Hot Flash Score (HFS) [Elkins et al. 2013], calculated through daily measurements as follows: HFS = frequency × average severity of hot flashes, where severity is rated from 1 to 4 (1: mild, 2: moderate, 3: severe, 4: very severe). The weekly HFS is calculated by averaging the daily HFS scores for each patient.
  Secondly, we will also evaluate the effect of guided self-hypnosis in reducing the frequency of hot flashes.

SECONDARY OUTCOMES:
Patient adherence | 28 days
  calculated from the data automatically recorded by the digital solution software. Adherence is thus evaluated by the rate of session follow-ups, estimated by the proportion of patients who followed all the recommended sessions without interruption, for the hypnosis group only.
Score of quality of life | 28 days
  Assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire at Day 0 and Day 28. The global score ranges from 0 to 100. For each question the scale ranges from 0 = not at all to 4 = a lot.
Sleep quality | 28 days
  Evaluated using the Pittsburgh Sleep Quality Index questionnaire score at Day 0 and Day 28. The global score ranges from 0 to 21. Higher scores indicate poorer sleep quality, with a score greater than 5 suggesting significant sleep difficulties.
Patient satisfaction | 28 days
  Assessed at Day 28 using a numerical scale. The numerical scale ranges from 0 = not satisfied to 10 = very satisfied.
Usability of the digital tool | 28 days
  Assessed at Day 28 using the System Usability Scale questionnaire score (Gronier & Baudet, 2021) for the hypnosis group only. It's composed of 10 questions on a scale from 0 = strongly disagree to 5 = strongly agree

CONTACTS AND LOCATIONS:
Overall Officials: AURELIEN LAMBERT, MD, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy, France